CLINICAL TRIAL: NCT01748747
Title: Peptide Vaccine With Resiquimod as an Immune Modulator for Patients With Resected Melanoma: A Pilot Study
Brief Title: Vaccine Therapy and Resiquimod in Treating Patients With Stage II-IV Melanoma That Has Been Removed By Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC0972; NCI-2012-01610 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Recurrent Melanoma; Stage IIA Melanoma; Stage IIB Melanoma; Stage IIC Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51; MART-1 Antigen; resiquimod; S 28463

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (MART-1 antigen, Gag:267-274 peptide vaccine) (Experimental): Patients receive MART-1 antigen and Gag:267-274 peptide vaccine emulsified in Montanide ISA 51 VG SC on day 1.
  Interventions: Drug: Montanide ISA 51 VG; Biological: MART-1 antigen; Other: laboratory biomarker analysis; Biological: Gag:267-274 peptide vaccine
- Arm II (MART-1 antigen, resiquimod, Montanide ISA 51 VG) (Experimental): Patients receive MART-1 antigen emulsified in Montanide ISA 51 VG SC followed by resiquimod applied topically on day 1.
  Interventions: Drug: Montanide ISA 51 VG; Biological: MART-1 antigen; Other: laboratory biomarker analysis
- Arm III (MART-1 antigen, Gag:267-274 peptide, resiquimod) (Experimental): Patients receive MART-1 antigen and Gag:267-274 peptide vaccine peptide vaccine emulsified in Montanide ISA 51 VG SC followed by resiquimod applied topically on day 1.
  Interventions: Drug: Montanide ISA 51 VG; Biological: MART-1 antigen; Other: laboratory biomarker analysis; Biological: Gag:267-274 peptide vaccine; Drug: resiquimod

INTERVENTIONS:
Drug: Montanide ISA 51 VG — Given SC
Biological: MART-1 antigen — Given SC
  Other Names: Antigen LB39-AA; Antigen SK29-AA; MART-1; MART-1 Tumor Antigen
Other: laboratory biomarker analysis — Correlative studies
Biological: Gag:267-274 peptide vaccine — Given SC
  Other Names: ILGLNKIV
  Arms: Arm I (MART-1 antigen, Gag:267-274 peptide vaccine); Arm III (MART-1 antigen, Gag:267-274 peptide, resiquimod)
Drug: resiquimod — Applied topically
  Other Names: R 848; S 28463
  Arms: Arm III (MART-1 antigen, Gag:267-274 peptide, resiquimod)

SUMMARY:
This pilot clinical trial studies vaccine therapy and resiquimod in treating patients with stage II-IV melanoma that has been removed by surgery. Vaccines made from peptides may help the body build an effective immune response to kill tumor cell tumor cells. Biological therapies, such as resiquimod, may stimulate the immune system in different ways and stop tumor cells from growing. It is not yet known whether Gag:267-274 peptide vaccine and resiquimod are more effective when given together or separately

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the immune response of each immunization regimen and determine an optimal regimen in terms of immune response to recommend for phase II testing.

SECONDARY OBJECTIVES:

I. Evaluate the adverse events profile of each immunization regimen. II. Evaluate disease-free survival.

TERTIARY OBJECTIVES:

I. Describe the immunological efficacy of the vaccine preparations with Gag267-274 (Gag:267-274 peptide vaccine) and resiquimod, as measured by the frequency and interferon (IFN)gamma production of peptide-specific cytotoxic T lymphocytes (CTL).

II. Examine immune responses to the tumor antigen analog MART-1a (MART-1 antigen) versus the xenoantigen Gag267-274.

OUTLINE: Patients are assigned to 1 of 3 treatment groups.

ARM I: Patients receive MART-1 antigen and Gag:267-274 peptide vaccine emulsified in Montanide ISA 51 VG subcutaneously (SC) on day 1.

ARM II: Patients receive MART-1 antigen emulsified in Montanide ISA 51 VG SC followed by resiquimod applied topically on day 1.

ARM III: Patients receive MART-1 antigen and Gag:267-274 peptide vaccine emulsified in Montanide ISA 51 VG SC followed by resiquimod applied topically on day 1.

In all arms, treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 9, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Central pathology review submission; this review for MART-1 positivity is mandatory prior to registration to confirm eligibility
* Human leukocyte antigen (HLA)-A2-positive
* Histologic proof of stage II, III or IV melanoma that has been completely resected with no current evidence of disease, as demonstrated by imaging within 2 months (stage III or stage IV; must be computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography [PET]/CT) or 6 months (stage II; may be chest x-ray, CT, MRI, or PET/CT)
* Absolute neutrophil count (ANC) >= 1500 mL
* Hemoglobin (Hgb) > 10 g/dL
* Platelets (PLT) >= 50,000 mL
* Aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Alkaline phosphatase =< 3 x ULN
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* For women of childbearing potential, a negative serum pregnancy test =< 7 days prior to registration
* Willingness to provide mandatory blood samples for correlative research

Exclusion Criteria:

* Uncontrolled or current infection
* Known standard therapy for the patient's disease that is potentially curative or proven capable of extending life expectancy
* Known allergy to vaccine or adjuvant components
* Any of the following prior therapies with interval since most recent treatment:

  * Chemotherapy =< 4 weeks prior to registration
  * Biologic therapy or immunotherapy =< 4 weeks prior to registration
  * Radiation therapy =< 4 weeks prior to registration
* Failure to fully recover from side effects of prior chemotherapy or surgery
* Any of the following, as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* Known immune deficiency, including human immunodeficiency virus (HIV) infection, as patients with known immune deficiencies will likely not be able to mount an immune response to the study vaccine; in addition, study patients should be naive to the HIV-derived Gag267-274 antigen
* History of systemic autoimmune disease, as patients with ongoing autoimmunity may be at an increased risk of autoimmune toxicity from the study vaccine
* Current or recent (=< 4 weeks prior to registration) use of immunosuppressive medications including systemic corticosteroids; (use of corticosteroids in doses not exceeding those used for adrenal replacement is acceptable)
* History of brain metastases (even if completely resected)
* Other active malignancy =< 5 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, they must not be receiving other treatment for their cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-12-14 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Immune response of each vaccination regimen, defined as a 2-fold or more increase from pre-treatment levels in the frequency of vaccine peptide-specific CTL as measured by tetramer staining | Up to 12 months
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true immune response rate will be calculated.

SECONDARY OUTCOMES:
Disease-free survival | From registration to recurrence, new primary, or death due to any cause, assessed up to 24 months
  Estimated using the method of Kaplan-Meier.
Incidence of adverse events, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 24 months
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States